CLINICAL TRIAL: NCT02554331
Title: Recherche et Mesure d'Anomalies précoces de la Marche au Cours Des Troubles du Comportement en Sommeil Paradoxal Idiopathiques
Brief Title: Gait and REM Sleep Behavior Disorder
Acronym: RBD-M2H
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9183
Record Dates: First submitted 2015-05-06; First posted 2015-09-18 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease; REM Sleep Behavior Disorder
Keywords: Gait; REM sleep behavior disorder; Parkinson's disease; Follow-up
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients RBD (Experimental): Patients RBD subject to FP-CIT single-photon emission computed tomography and Neuropsychological evaluation and Gait recording with sensors
  Interventions: Radiation: FP-CIT single-photon emission computed tomography; Behavioral: neuropsychological evaluation; Other: Gait recording with sensors
- controls healthy volunteers (Other): controls healthy volunteers subject to Neuropsychological evaluation and Gait recording with sensors
  Interventions: Behavioral: neuropsychological evaluation; Other: Gait recording with sensors

INTERVENTIONS:
Radiation: FP-CIT single-photon emission computed tomography — FP-CIT radiolabeled is used as a surrogate marker to examine the integrity of the dopaminergic nigrostriatal neurons.
  Arms: Patients RBD
Behavioral: neuropsychological evaluation — Assessment of:
  * overall cognitive function
  * executive functions
  * visuospatial functions
  * Nonverbal memory
  * verbal memory
  * Evaluation of hearing ability of time perception and sensorimotor synchronization from selected tasks the Battery of assessment of auditory sensorimotor and timing abilities
  * Beck Depression Inventory
Other: Gait recording with sensors — Gait recording with sensors

SUMMARY:
Many people with idiopathic rapid eye movement (REM) sleep behavior disorder (RBD) have an underlying synucleinopathy, the most common of which are Parkinson's disease (PD) and Lewy body disease. Identifying additional abnormal clinical features may help in identifying those at greater risk of evolving to a more severe syndrome. Because gait disorders are common in the synucleinopathies, early abnormalities in gait in those with RBD could help in identifying those at increased risk of developing overt parkinsonism and/or cognitive impairment.

The investigators aim to identify subtle gait abnormalities in idiopathic RBD and to identify sensitive and early biomarkers:

1. to detect subtle gait disorders in pre-symptomatic stage of synucleinopathy and
2. to track their evolution in the parallel with the disease progression.

Main objective: In comparison with age and gender matched-controls, to identify in patients with RBD a larger reduction of gait velocity (and other abnormalities of spatio-temporal characteristics of gait) between a single (gait) and a dual-task (gait+cognitive task).

Secondary objective:

1. In comparison with age and gender matched-PD patients, to identify in patients with RBD a smaller reduction of gait velocity (and other abnormalities of spatio-temporal characteristics of gait) between a single (gait) and a dual-task (gait+cognitive task).
2. In patients with RBD to identify correlations between the spatio-temporal characteristics modifications of gait between a single (gait) and a dual-task (gait+cognitive task) and the percentage of REM without atonia - the dopamine transporter (DAT) density using FP-CIT single-photon emission computed tomography; the reduction of the olfactory discrimination and thresholds.
3. In patients with RBD to track the spatio-temporal characteristics evolution of gait over time (every 6 months for 2 years)

ELIGIBILITY:
Inclusion Criteria:

* Specific inclusion criteria for RBD patients - to reach the diagnosis criteria of RBD (International Classification of Sleep Disorders 2)
* Specific inclusion criteria for PD patients - to reach the diagnosis criteria of idiopathic PD (Queen Square Brain Bank) - Hoehn Yahr score ≤ 2

Exclusion Criteria:

* Specific exclusion criteria for RBD patients - diagnosis of PD - other pathology associated to RBD diagnosis - presence of antiparkinsonism medication
* Specific exclusion criteria for PD patients - clinical signs of parkinsonian syndrome- Mini Mental State Examination < 24/30- gait disorder clinically observable
* Specific exclusion criteria for controls - neurological disease- gait disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2015-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
gait velocity | Month 24
  gait speed difference between single and dual tasks

SECONDARY OUTCOMES:
spatio-temporal gait characteristics | Month 24
  oscillation phase duration difference between single and dual tasks

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Cochen De Cock, MD, Principal Investigator — University Hospital
Locations (1):
- University hospital, Montpellier, France